CLINICAL TRIAL: NCT01342848
Title: REduction of Myocardial Necrosis Achieved With Nose-dive Manual Thrombus Aspiration
Brief Title: Effectiveness of Thrombus Aspiration in Plaque Reduction for Patients With Acute Coronary Syndromes
Acronym: REMNANT
Status: Completed | Type: Observational
Sponsor: Raffaele De Caterina (Other)
Collaborators: San Giovanni Addolorata Hospital (Other)
Responsible Party: Sponsor-Investigator, Raffaele De Caterina, Director - Institute of Cardiology, G. d'Annunzio University
Organization: G. d'Annunzio University (Other)
Other Study IDs: 2010-021835-15
Record Dates: First submitted 2011-04-12; First posted 2011-04-27 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Acute Coronary Syndrome
Keywords: NSTE-ACS; PCI; Thrombus Aspiration; IVUS; Periprocedural Myocardial Infarction
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — Histopathology assessment of aspirated material during manual TA. Quantitative analysis: size and weight. Qualitative evaluation: a) thrombus containing only platelets, b) a thrombus with an erythrocyte component c) any fragment of vessel wall, cholesterol crystals, inflammatory cells or collagen tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Although successful, percutaneous coronary interventions (PCI) with stent implantation may be hampered by periprocedural myocardial necrosis. In acute ST-elevation myocardial infarction (STEMI), the reduction of thrombus burden through manual thrombus aspiration (TA) of an occluded coronary artery has been documented to produce an improved myocardial perfusion rate and significant survival advantage. To date, beyond feasibility and safety studies no clinical benefit has been yet documented with the use of TA before stent deployment in the setting of acute coronary syndromes (ACS) outside acute STEMI. The investigators hypothesize that TA before stent deployment reduces the thrombus/plaque burden - as assessed by intravascular imaging systems - in the setting of acute coronary syndromes (ACS) outside acute STEMI.

DETAILED DESCRIPTION:
Periprocedural myocardial infarction (MI) has an independent adverse prognostic relevance. Several trials have documented a reduction in the occurrence of periprocedural MI through various pharmacological strategies, with enhanced inhibition of platelet aggregation or high dose statins. However, real-world registries still document an incidence of periprocedural MI in 30-40% of patients. Currently available intravascular imaging techniques, Intravascular Ultrasound (IVUS) and more recently available Optical Coherence Tomography (OCT) allow a precise evaluation of the coronary plaque and can be extremely useful for monitoring plaque modifications obtained with thrombus aspiration (TA). Plaque burden will be assessed as plaque + media (P+M), commonly measured with IVUS by subtracting lumen (L) to external elastic membrane (EEM) cross sectional area (P+M= EEM-L).

Expecting a mean plaque volume of 160±50 mm3 in a population of patients with ACS undergoing PCI, a sample size of at least 45 patients (52 lesions) with a recent (<15 days, but after 24 hours) STEMI or a non-ST elevation (NSTE)-ACS within 72 hours of symptoms would provide a 90% power to detect a 20% reduction in the plaque volume after TA with an alpha (probability value) of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75 years old.
* Recent(<15 days, >24 hrs)STEMI or NSTE-ACS within 72 hrs of symptoms.
* Presence at least one "culprit" high-grade (>90%)lesion.

Exclusion Criteria:

* STEMI within 24 hours.
* Cardiogenic shock, decompensated heart failure, LVEF<30%.
* Serum creatinine ≥ 2.5 mg/dl.
* Contraindication to aspirin, heparin, thienopyridines.
* Total occlusion of target vessel.
* Diseased vein graft or a restenosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 patients with at least one "culprit" lesion, identified as a high-grade (>90%) lesion in the territory of jeopardized myocardium, at coronary angiography performed for a recent (<15 days, but after 24 hours) STEMI or a non-ST elevation (NSTE)-ACS within 72 hours of symptoms.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The change in plaque volume as assessed by intravascular ultrasound (IVUS). | From baseline to 10 minutes after thromboaspiration (TA)
  The reduction of plaque volume after TA, assessed as (Baseline P+M)- (Post-TA P+M);

SECONDARY OUTCOMES:
Histopathology assessment of aspirated material. | One week after PCI
  Quantitative analysis: size and weight. Qualitative evaluation: a) thrombus containing only platelets, b) a thrombus with an erythrocyte component c) any fragment of vessel wall, cholesterol crystals, inflammatory cells or collagen tissue.
Myocardial infarct size by markers of myocardial injury/necrosis | Up to 72 hours after PCI
  Myocardial infarct size will be determined as the area under the curve of serial CK-MB and cardiac Troponin I assessment
The change in thrombus burden as assessed by Optical Coherence Tomography (OCT) | From baseline to 10 minutes after thromboaspiration (TA)
  Thrombus burden will be assessed with a semiquantitative scale (0-4) by OCT at baseline and after TA

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Center of Predictive Molecular Medicine - University "G. d'Annunzio", Chieti
  - Institute of Cardiology, G. d'Annunzio University, Chieti
  - San Giovanni Hospital and Centro per la Lotta Contro l'Infarto, Fondazione Onlus, Rome

REFERENCES:
- [Background] Silber S, Albertsson P, Aviles FF, Camici PG, Colombo A, Hamm C, Jorgensen E, Marco J, Nordrehaug JE, Ruzyllo W, Urban P, Stone GW, Wijns W; Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Guidelines for percutaneous coronary interventions. The Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Eur Heart J. 2005 Apr;26(8):804-47. doi: 10.1093/eurheartj/ehi138. Epub 2005 Mar 15. PMID 15769784
- [Background] Iakovou I, Mintz GS, Dangas G, Abizaid A, Mehran R, Kobayashi Y, Lansky AJ, Aymong ED, Nikolsky E, Stone GW, Moses JW, Leon MB. Increased CK-MB release is a "trade-off" for optimal stent implantation: an intravascular ultrasound study. J Am Coll Cardiol. 2003 Dec 3;42(11):1900-5. doi: 10.1016/j.jacc.2003.06.012. PMID 14662249
- [Background] Prati F, Pawlowski T, Gil R, Labellarte A, Gziut A, Caradonna E, Manzoli A, Pappalardo A, Burzotta F, Boccanelli A. Stenting of culprit lesions in unstable angina leads to a marked reduction in plaque burden: a major role of plaque embolization? A serial intravascular ultrasound study. Circulation. 2003 May 13;107(18):2320-5. doi: 10.1161/01.CIR.0000066695.24697.07. Epub 2003 Apr 21. PMID 12707236
- [Background] Nienhuis MB, Ottervanger JP, Bilo HJ, Dikkeschei BD, Zijlstra F. Prognostic value of troponin after elective percutaneous coronary intervention: A meta-analysis. Catheter Cardiovasc Interv. 2008 Feb 15;71(3):318-24. doi: 10.1002/ccd.21345. PMID 18288753
- [Background] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction. Universal definition of myocardial infarction. Eur Heart J. 2007 Oct;28(20):2525-38. doi: 10.1093/eurheartj/ehm355. No abstract available. PMID 17951287
- [Background] Kastrati A, Mehilli J, Neumann FJ, Dotzer F, ten Berg J, Bollwein H, Graf I, Ibrahim M, Pache J, Seyfarth M, Schuhlen H, Dirschinger J, Berger PB, Schomig A; Intracoronary Stenting and Antithrombotic: Regimen Rapid Early Action for Coronary Treatment 2 (ISAR-REACT 2) Trial Investigators. Abciximab in patients with acute coronary syndromes undergoing percutaneous coronary intervention after clopidogrel pretreatment: the ISAR-REACT 2 randomized trial. JAMA. 2006 Apr 5;295(13):1531-8. doi: 10.1001/jama.295.13.joc60034. Epub 2006 Mar 13. PMID 16533938
- [Background] Patti G, Colonna G, Pasceri V, Pepe LL, Montinaro A, Di Sciascio G. Randomized trial of high loading dose of clopidogrel for reduction of periprocedural myocardial infarction in patients undergoing coronary intervention: results from the ARMYDA-2 (Antiplatelet therapy for Reduction of MYocardial Damage during Angioplasty) study. Circulation. 2005 Apr 26;111(16):2099-106. doi: 10.1161/01.CIR.0000161383.06692.D4. Epub 2005 Mar 6. PMID 15750189
- [Background] Pasceri V, Patti G, Nusca A, Pristipino C, Richichi G, Di Sciascio G; ARMYDA Investigators. Randomized trial of atorvastatin for reduction of myocardial damage during coronary intervention: results from the ARMYDA (Atorvastatin for Reduction of MYocardial Damage during Angioplasty) study. Circulation. 2004 Aug 10;110(6):674-8. doi: 10.1161/01.CIR.0000137828.06205.87. Epub 2004 Jul 26. PMID 15277322
- [Background] Svilaas T, Vlaar PJ, van der Horst IC, Diercks GF, de Smet BJ, van den Heuvel AF, Anthonio RL, Jessurun GA, Tan ES, Suurmeijer AJ, Zijlstra F. Thrombus aspiration during primary percutaneous coronary intervention. N Engl J Med. 2008 Feb 7;358(6):557-67. doi: 10.1056/NEJMoa0706416. PMID 18256391
- [Background] Vlaar PJ, Diercks GF, Svilaas T, Vogelzang M, de Smet BJ, van den Heuvel AF, Anthonio RL, Jessurun GA, Tan ES, Suurmeijer AJ, Zijlstra F. The feasibility and safety of routine thrombus aspiration in patients with non-ST-elevation myocardial infarction. Catheter Cardiovasc Interv. 2008 Dec 1;72(7):937-42. doi: 10.1002/ccd.21717. PMID 19021272
- [Background] Zimarino M, Prati F, Stabile E, Pizzicannella J, Fouad T, Filippini A, Rabozzi R, Trubiani O, Pizzicannella G, De Caterina R. Optical coherence tomography accurately identifies intermediate atherosclerotic lesions--an in vivo evaluation in the rabbit carotid artery. Atherosclerosis. 2007 Jul;193(1):94-101. doi: 10.1016/j.atherosclerosis.2006.08.047. Epub 2006 Sep 27. PMID 17007862
- [Background] Prati F, Regar E, Mintz GS, Arbustini E, Di Mario C, Jang IK, Akasaka T, Costa M, Guagliumi G, Grube E, Ozaki Y, Pinto F, Serruys PW; Expert's OCT Review Document. Expert review document on methodology, terminology, and clinical applications of optical coherence tomography: physical principles, methodology of image acquisition, and clinical application for assessment of coronary arteries and atherosclerosis. Eur Heart J. 2010 Feb;31(4):401-15. doi: 10.1093/eurheartj/ehp433. Epub 2009 Nov 4. PMID 19892716
- [Background] Naghavi M, Libby P, Falk E, Casscells SW, Litovsky S, Rumberger J, Badimon JJ, Stefanadis C, Moreno P, Pasterkamp G, Fayad Z, Stone PH, Waxman S, Raggi P, Madjid M, Zarrabi A, Burke A, Yuan C, Fitzgerald PJ, Siscovick DS, de Korte CL, Aikawa M, Juhani Airaksinen KE, Assmann G, Becker CR, Chesebro JH, Farb A, Galis ZS, Jackson C, Jang IK, Koenig W, Lodder RA, March K, Demirovic J, Navab M, Priori SG, Rekhter MD, Bahr R, Grundy SM, Mehran R, Colombo A, Boerwinkle E, Ballantyne C, Insull W Jr, Schwartz RS, Vogel R, Serruys PW, Hansson GK, Faxon DP, Kaul S, Drexler H, Greenland P, Muller JE, Virmani R, Ridker PM, Zipes DP, Shah PK, Willerson JT. From vulnerable plaque to vulnerable patient: a call for new definitions and risk assessment strategies: Part I. Circulation. 2003 Oct 7;108(14):1664-72. doi: 10.1161/01.CIR.0000087480.94275.97. PMID 14530185
- [Background] Zimarino M, Calafiore AM, De Caterina R. Complete myocardial revascularization: between myth and reality. Eur Heart J. 2005 Sep;26(18):1824-30. doi: 10.1093/eurheartj/ehi249. Epub 2005 Apr 11. PMID 15824076